CLINICAL TRIAL: NCT05076253
Title: Efficacy and Safety of Ivermectin in Treatment of Mild to Moderate COVID-19 Infection: a Randomized ,Double Blind,Placebo,Controlled Trial
Brief Title: Efficacy of Ivermectin in COVID-19
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Bangkok Metropolitan Administration Medical College and Vajira Hospital (Other Government)
Responsible Party: Principal Investigator, Thananda Trakarnvanich, Associate Professor, Bangkok Metropolitan Administration Medical College and Vajira Hospital
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: 171/64
Record Dates: First submitted 2021-10-08; First posted 2021-10-13 (Actual); Last update posted 2021-12-15 (Actual); Status verified 2021-12

CONDITIONS: Safety; SARS-CoV2 Infection; Ivermectin Poisoning; Effect of Drug
Keywords: efficacy; ivermectin; covid-19; randomised controlled trial
MeSH Terms: conditions — COVID-19 | interventions — Ivermectin

STUDY DESIGN:
Intervention Model Description: a randomized ,double blind,placebo,controlled trial
Who Masked: Participant, Care Provider, Investigator
Masking Description: Group A: Ivermectin Group B: Placebo
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ivermectin (Active Comparator): Ivermectin 12 mg per day for 5 plus standard care
  Interventions: Drug: Ivermectin; Drug: Placebo
- Placebo (Placebo Comparator): Placebo plus standard care
  Interventions: Drug: Ivermectin; Drug: Placebo

INTERVENTIONS:
Drug: Ivermectin — Ivermectin plus standard care
Drug: Placebo — Standard care

SUMMARY:
The newly emerged corona virus disease 2019 (COVID-19) has spread to all over the world, with recent estimates of more than 236 million cases diagnosed and led to 4.8 million deaths as November 20211 .Therapeutic approaches are needed to improve outcomes in patients with COVID-19 since no antiviral agent has yet been proved to be conclusively beneficial in COVID-19 infection,especially in patients with mild to moderate degree of severity There has been growing interest in the anti-parasitic drug,ivermectin, which previously was studied as an antiviral, anti-inflammatory and anti-cancer actions2 .It was also reported to have an in-vitro activity against SARS-CoV-23 .Its antiviral properties was due to the action on importin 2/1 mediated nuclear transport. Ivermectin prevents the binding of viral proteins to importin 2/1 rendering the viral proteins unable to enter the nucleus and cause infection4.

Several clinical studies have found a beneficial effect of ivermectin in COVID-195-9 However, some study did not find significant difference between the patient group receiving ivermectin and control group10 .Until now, the controlled trials evaluating ivermectin in COVID-19 are lacking. Ivermectin is safe, with reported side effect of less than 1%. Hence it is essential to conduct a clinical trial with ivermectin in patients with COVID-19 .The objective of this study is to establish the efficacy of ivermectin for COVID-19 patients with mild to moderate disease, compare to usual case alone.

DETAILED DESCRIPTION:
This study is a randomized, double-blind, placebo controlled trial conducted at Faculty of Medicine, Vajira Hospital, Navamindradhiraj University from September 2021 to the end of November 2021.

The patients were randomized in permuted block of four in a randomized sequence prepared by the unblinded pharmacist in Microsoft excel12 .Allocation assignment was concealed from investigators and the patients. The patients were allocated into two groups : either to group A (Ivermectin arm) or to group B (control arm) as shown in Fig 1. The patients were randomized in a 1:1 ratio .Group A received ivermectin 12 mg per day for 5 days as recommended by previous studes13,14 plus standard care. Group B was to receive standard care alone which included favipiravir or andrographolide, corticosteroids, cetrizine and paracetamol.

ELIGIBILITY:
Inclusion Criteria:

* adult men and women age 18-80 years
* non-pregnant or breast-feeding women
* had mild to moderate symptoms as defined by the World Health Organization (WHO) severity score for COVID-19 Mild disease was defined as cough , runny nose,anosmia, fever, diarrhea without dyspnea or tachypnea.

Moderate disease was defined as pneumonia but with oxygen saturation more than 90 percent

Exclusion Criteria:

* were allergic to ivermectin
* have the potential for a drug-drug interaction with ivermectin such as tamoxifen or warfarin
* previously treated with ivermectin in the last 7 days
* had received any herbal medicine
* had severe chronic illness (severe congestive heart failure, chronic kidney disease stage 4-5, chronic liver disease, terminal cancer diseases)
* had concurrent bacterial infection or unwilling to participate in the trial
* Patients with severe symptoms, likely due to cytokine release syndrome
* uncontrolled co-morbidities and immunocompromised states

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 72 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Viral clearance of SARS- CoV-2 intervention | 7 days
  Viral load from RT-PCR test
Viral clearance of SARS- CoV-2 intervention | 14 days
  Viral load from RT-PCR test

SECONDARY OUTCOMES:
Duration of hospitalization | 28 days
  Day of hospitalization
frequency of clinical worsening | 28 days
  numbers of cases that have clinical worsening
Mechanical ventilation | 28 days
  numbers of cases that needs mechanical ventilation
Mortality rate | 28 days
  numbers of cases that died

CONTACTS AND LOCATIONS:
Overall Officials: Thananda Trakarnvanich, M.D., Principal Investigator — Bangkok Metropolitan Administration and Vajira Hospital
Locations (1):
- Thananda Trakarnvanich, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Yes
Data will be made available upon request after publication
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After publication

REFERENCES:
- [Background] Omura S, Crump A. Ivermectin: panacea for resource-poor communities? Trends Parasitol. 2014 Sep;30(9):445-55. doi: 10.1016/j.pt.2014.07.005. Epub 2014 Aug 12. PMID 25130507
- [Background] Chen IS, Kubo Y. Ivermectin and its target molecules: shared and unique modulation mechanisms of ion channels and receptors by ivermectin. J Physiol. 2018 May 15;596(10):1833-1845. doi: 10.1113/JP275236. Epub 2017 Nov 9. PMID 29063617
- [Background] Khan MSI, Khan MSI, Debnath CR, Nath PN, Mahtab MA, Nabeka H, Matsuda S, Akbar SMF. Ivermectin Treatment May Improve the Prognosis of Patients With COVID-19. Arch Bronconeumol (Engl Ed). 2020 Dec;56(12):828-830. doi: 10.1016/j.arbres.2020.08.007. Epub 2020 Sep 24. No abstract available. PMID 33293006
- [Background] Ahmed S, Karim MM, Ross AG, Hossain MS, Clemens JD, Sumiya MK, Phru CS, Rahman M, Zaman K, Somani J, Yasmin R, Hasnat MA, Kabir A, Aziz AB, Khan WA. A five-day course of ivermectin for the treatment of COVID-19 may reduce the duration of illness. Int J Infect Dis. 2021 Feb;103:214-216. doi: 10.1016/j.ijid.2020.11.191. Epub 2020 Dec 2. PMID 33278625
- [Derived] Manomaipiboon A, Pholtawornkulchai K, Poopipatpab S, Suraamornkul S, Maneerit J, Ruksakul W, Phumisantiphong U, Trakarnvanich T. Efficacy and safety of ivermectin in the treatment of mild to moderate COVID-19 infection: a randomized, double-blind, placebo-controlled trial. Trials. 2022 Aug 26;23(1):714. doi: 10.1186/s13063-022-06649-3. PMID 36028897